CLINICAL TRIAL: NCT03663868
Title: Cumulus Cell mRNA Analysis as Oocyte Quality Marker in the Fertility Lab in a Prospective Single-center Study for rFSH Stimulated Patients
Brief Title: Single-center Prospective Cumulus Cell Test Study in rFSH Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BUN143201318000 b
Record Dates: First submitted 2018-09-03; First posted 2018-09-10 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CC-Test diagnosis and Day 3 transfer (Experimental): Patients undergo the standard ART treatment, as described by the treating physician, with standard morphology based scoring of the embryos + the extra cumulus cell based diagnosis and transfer of the best embryo based on morphology and CC diagnosis on day 3 of embryo growth (cleavage stage embryo)
  Interventions: Diagnostic Test: CC-Test
- Day 3 transfer control group (No Intervention): Patients undergo the standard ART treatment, as described by the treating physician, with standard morphology based scoring of the embryos and transfer of the best embryo based on morphology on day 3 of embryo growth (cleavage stage embryo)
- Day 5 transfer control group (No Intervention): Patients undergo the standard ART treatment, as described by the treating physician, with standard morphology based scoring of the embryos and transfer of the best embryo based on morphology on day 5 of embryo growth (blastocyst stage embryo)

INTERVENTIONS:
Diagnostic Test: CC-Test — Classification of the oocyte/embryo based on the gene expression pattern observed in the cumulus cells
  Arms: CC-Test diagnosis and Day 3 transfer

SUMMARY:
Performing an additional non-invasive oocyte diagnostic test based on cumulus cell gene expression could improve the outcome of the ART cycle for rFSH stimulated patients

ELIGIBILITY:
Inclusion Criteria:

* scheduled for intracytoplasmatic sperm injection (ICSI) and single (or double) embryo transfer on day 3
* patients down regulated with gonadotropin-releasing hormone (GnRH) antagonist and stimulated with recombinant Follicle Stimulating Hormone (FSH)
* undergoing first or second IVF or ICSI cycle with transfer
* Body Mass Index (BMI) between 17 and 33
* regular menstrual cycle (between 24 and 35 days)

Exclusion Criteria:

* smokers (> 10 cigarettes per day)
* patients requesting Pre-implantation Genetic Diagnosis (PGD)
* patients with polycystic ovary syndrome (PCOS), or severe endometriosis (AFS stage 3-4)
* couples where the partner has an extremely low sperm count i.e.: extreme oligo-astheno-teratozoospermia (OAT) (< 100.000/ml) or scheduled for testicular sperm extraction (TESE)
* results of eventual preceding cycles may not indicate a known genetic disease, or low ovarian response or an oocyte maturation defect

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-14 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy as observed by ultrasound | 2 months after embryo transfer
  This observation is routinely performed by the treating physician for every patient undergoing standard ART treatment and is thus available from the fertility center database

SECONDARY OUTCOMES:
Positive beta-hCG pregnancy as observed by serum analysis | 12-17 days after embryo transfer
  This observation is routinely performed by the treating physician for every patient undergoing standard ART treatment and is thus available from the fertility center database
Live birth by questionnaire | at least 9 months after embryo transfer
  This observation is routinely performed by the study nurses of the fertility center for every patient undergoing standard ART treatment and is thus available from the fertility center database. This measurement does not include a scale, there is either a child born or not. The date of delivery and the gender of the child are asked together with eventual complications.
Cumulative pregnancy by ultrasound (for pregnancy follow-up) and questionnaire (for live birth follow-up) (see outcome 1 and 3) | 2 years after embryo transfer
  This is the compilation of the data gathered in outcome 1 and 3 for eventual consecutive cycles. This observation is routinely performed by the study nurses of the fertility center for every patient undergoing standard ART treatment and is thus available from the fertility center database

CONTACTS AND LOCATIONS:
Overall Officials: Johan Smitz, Prof. Dr., Study Director — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No